CLINICAL TRIAL: NCT05689957
Title: Evaluation of Surgical Condition During Laparoscopic Gynaecological Surgery in Patient With Moderate vs Deep Neuromuscular Block in Lower Pressure Pneumoperitoneum
Brief Title: Moderate vs Deep Neuromuscular Block in Lower Pressure Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Profesor Madya Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USM/JEPeM/20080410
Record Dates: First submitted 2020-12-30; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Disease; Neuromuscular Blockade
Keywords: deep neuromuscular block; low pressure pneumoperitoneum; laparoscopic gynaecological surgery
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- deep neuromuscular block group (Experimental): Group 1 (Induction with Rocuronium 0.6mg/kg + maintenance with intravenous Rocuronium rocuronium 8-12mcg/kg/minute (0.48-0.72 mg/kg/hour maintain PTC 0-1(deep block). (Study Group) intraoperatively
  Interventions: Drug: Deep neuromuscular block using intravenous rocuronium induction at 1.2mg/kg and maintainance of 8-12mcg/kg/min for deep neuromuscular block
- moderate neuromuscular block group (Active Comparator): Group 2 (Induction with intravenous Rocuronium 0.6mg/kg + maintenance with intermittent intravenous Rocuronium 0.2mg/kg bolus. maintain PTC >1, TOF 0-2). Moderate block. (Control Group) intraoperatively
  Interventions: Drug: Deep neuromuscular block using intravenous rocuronium induction at 1.2mg/kg and maintainance of 8-12mcg/kg/min for deep neuromuscular block

INTERVENTIONS:
Drug: Deep neuromuscular block using intravenous rocuronium induction at 1.2mg/kg and maintainance of 8-12mcg/kg/min for deep neuromuscular block — both arm are using low pressure pneumoperitoneum in laparoscopic surgery, moderate and deep neuromuscular block are monitor with neuromuscular monitoring. if surgical condition is inadequate, surgeon are allowed to increase intraabdominal pressure as per standard care

SUMMARY:
The investigators hypothesized that deep neuromuscular block compare to moderate neuromuscular block would reduce the rate of increasing intraabdominal pressure and operation can be completely done in lower pressure pneumoperitoneum and would improve laparoscopic space by measuring distance from the sacral promontory to the inserted trocar in patients undergoing laparoscopic gynaecological surgery.

DETAILED DESCRIPTION:
Laparoscopic surgery has increasing popularity and slowly replacing conventional open surgery as it offers more benefit to patient and health care practitioner. The overall risk of complications during laparoscopic surgery is recognized to be lower than during laparotomy. Laparoscopic hysterectomy compare to open vaginal hysterectomy reduces postoperative pain, reduce post op analgesics requirement and shorter duration of hospital admission.1 However, the increase intra-abdominal pressure created during laparoscopic surgery can affect cardiovascular, pulmonary and renal physiology. Besides the risk of post-operative nausea and vomiting, it is also stated that the pneumoperitoneum created during laparoscopic surgery is an important factor in the cause of postoperative shoulder pain.2 Traditionally pneumoperitoneum created at 15mmHg3. Insufflation of intraabdominal carbon dioxide may cause post-operative shoulder pain up to 70% in some study in gynaecologic laparoscopic surgery. 4 Use a lower pressure pneumoperitoneum might decrease postoperative pain, decrease post-operative shoulder tip pain5 and reduce the risk of laparoscopic related complication6. Many studies used lower insufflation of intraabdominal pressure as an intraoperative intervention to reduce the complication7,8. However, a lower intraabdominal pressure may worsen surgical space and increase the risk of conversion to open surgery.

Though many factors contribute to the quality of surgical space include non-modifiable such as obesity, previous abdominal surgery and modifiable factors such as anaesthesia related factor, patient position and intraabdominal pressure. Numerous studies also have been carried out showing that deep neuromuscular block improves surgical condition in different type of laparoscopic surgery includes robotic assisted laparoscopic surgery.9,10,11 Currently with the advancement of technology where neuromuscular monitoring is widely available and the selective reversal binding agent suggamadex where post-operative complication of inadequate reversal can be markedly reduced, several studies have been done to observe the benefit of low intraabdominal pressure with deep neuromuscular block to surgical space quality and intraoperative complication related to high pressure intraabdominal complication compare to usual moderate block.9,10,12 However there is still few study objectively measure the possible effect of deep neuromuscular blocker on the surgical space and the ability of surgery to be completely done in low pressure pneumoperitoneum in laparoscopic gynaecological surgery.

This study will compare the rate of increasing intraabdominal pressure, skin to sacral promontary distance, and post operative pain between deep neuromuscular block and moderate neuromuscular block.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* ASA I or II
* schedule to undergo laparoscopic gynaecological surgery (laparoscopic hysterectomy and laparoscopic ovarian cystectomy in Hospital Universiti Sains Malaysia , Kubang Kerian, Kelantan

Exclusion Criteria:

* Allergy to study drugs (rocuronium, suggamadex)
* Serious cardiac and respiratory disease (reactive airway disease, upper respiratory tract infection)
* Neurological or neuromuscular disease (epilepsy, family history and history of malignant hyperthermia etc.)
* Pregnancy
* Morbid obesity BMI>35

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The adequacy of intraabdominal pressure in mmHg | intraoperative
  1. To compare the rate of increasing intra-abdominal pressure (IAP) by the surgeon when they decide that the surgical conditions are inadequate for the operation in patient receiving deep neuromuscular block compare to moderate neuromuscular block in laparoscopic gynaecological surgery

SECONDARY OUTCOMES:
The quality of surgical space | intraoperative
  2. To compare quality of surgical space condition in patient receiving deep and moderate neuromuscular block in laparoscopic gynaecological surgery.
the distance between the skin to sacral promontary in centimetres (cm) | intaoperative
  3. To compare skin to sacral promontory distance in patient in patient receiving moderate neuromuscular block and deep neuromuscular block in laparoscopic gynaecological surgery.
post operative pain | 24 hour post operation
  To compare the post-operative pain and shoulder tip pain in patient receiving deep neuromuscular block and moderate neuromuscular block in laparoscopic gynaecological surgery by using visual analog pain score (VAS)
shoulder tip pain using pain visual analogue score (VAS) | 24 hour post operation
  To compare shoulder tip pain in patient receiving deep neuromuscular block and moderate neuromuscular block in laparoscopic gynaecological surgery by using visual analog pain score (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Umairah Esa, MBBS, Principal Investigator
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Background] Ghezzi F, Uccella S, Cromi A, Siesto G, Serati M, Bogani G, Bolis P. Postoperative pain after laparoscopic and vaginal hysterectomy for benign gynecologic disease: a randomized trial. Am J Obstet Gynecol. 2010 Aug;203(2):118.e1-8. doi: 10.1016/j.ajog.2010.04.026. Epub 2010 Jun 3. PMID 20522410
- [Background] Madsen MV, Istre O, Staehr-Rye AK, Springborg HH, Rosenberg J, Lund J, Gatke MR. Postoperative shoulder pain after laparoscopic hysterectomy with deep neuromuscular blockade and low-pressure pneumoperitoneum: A randomised controlled trial. Eur J Anaesthesiol. 2016 May;33(5):341-7. doi: 10.1097/EJA.0000000000000360. PMID 26479510
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Background] Bogani G, Uccella S, Cromi A, Serati M, Casarin J, Pinelli C, Ghezzi F. Low vs standard pneumoperitoneum pressure during laparoscopic hysterectomy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):466-71. doi: 10.1016/j.jmig.2013.12.091. Epub 2013 Dec 25. PMID 24374246
- [Background] Kyle EB, Maheux-Lacroix S, Boutin A, Laberge PY, Lemyre M. Low vs Standard Pressures in Gynecologic Laparoscopy: a Systematic Review. JSLS. 2016 Jan-Mar;20(1):e2015.00113. doi: 10.4293/JSLS.2015.00113. PMID 26955258
- [Background] Donatsky AM, Bjerrum F, Gogenur I. Surgical techniques to minimize shoulder pain after laparoscopic cholecystectomy. A systematic review. Surg Endosc. 2013 Jul;27(7):2275-82. doi: 10.1007/s00464-012-2759-5. Epub 2013 Jan 24. PMID 23340814
- [Background] Kim MH, Lee KY, Lee KY, Min BS, Yoo YC. Maintaining Optimal Surgical Conditions With Low Insufflation Pressures is Possible With Deep Neuromuscular Blockade During Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-Blind, Parallel-Group Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2920. doi: 10.1097/MD.0000000000002920. PMID 26945393
- [Background] Koo BW, Oh AY, Seo KS, Han JW, Han HS, Yoon YS. Randomized Clinical Trial of Moderate Versus Deep Neuromuscular Block for Low-Pressure Pneumoperitoneum During Laparoscopic Cholecystectomy. World J Surg. 2016 Dec;40(12):2898-2903. doi: 10.1007/s00268-016-3633-8. PMID 27405749
- [Background] Madsen MV, Gatke MR, Springborg HH, Rosenberg J, Lund J, Istre O. Optimising abdominal space with deep neuromuscular blockade in gynaecologic laparoscopy--a randomised, blinded crossover study. Acta Anaesthesiol Scand. 2015 Apr;59(4):441-7. doi: 10.1111/aas.12493. Epub 2015 Mar 1. PMID 25789421
- [Background] Ozdemir-van Brunschot DMD, Braat AE, van der Jagt MFP, Scheffer GJ, Martini CH, Langenhuijsen JF, Dam RE, Huurman VA, Lam D, d'Ancona FC, Dahan A, Warle MC. Deep neuromuscular blockade improves surgical conditions during low-pressure pneumoperitoneum laparoscopic donor nephrectomy. Surg Endosc. 2018 Jan;32(1):245-251. doi: 10.1007/s00464-017-5670-2. Epub 2017 Jun 22. PMID 28643056
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Bruintjes MH, van Helden EV, Braat AE, Dahan A, Scheffer GJ, van Laarhoven CJ, Warle MC. Deep neuromuscular block to optimize surgical space conditions during laparoscopic surgery: a systematic review and meta-analysis. Br J Anaesth. 2017 Jun 1;118(6):834-842. doi: 10.1093/bja/aex116. PMID 28575335
- [Background] Park SK, Son YG, Yoo S, Lim T, Kim WH, Kim JT. Deep vs. moderate neuromuscular blockade during laparoscopic surgery: A systematic review and meta-analysis. Eur J Anaesthesiol. 2018 Nov;35(11):867-875. doi: 10.1097/EJA.0000000000000884. PMID 30188357
- [Background] Wei Y, Li J, Sun F, Zhang D, Li M, Zuo Y. Low intra-abdominal pressure and deep neuromuscular blockade laparoscopic surgery and surgical space conditions: A meta-analysis. Medicine (Baltimore). 2020 Feb;99(9):e19323. doi: 10.1097/MD.0000000000019323. PMID 32118762
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Background] Yoo YC, Kim NY, Shin S, Choi YD, Hong JH, Kim CY, Park H, Bai SJ. The Intraocular Pressure under Deep versus Moderate Neuromuscular Blockade during Low-Pressure Robot Assisted Laparoscopic Radical Prostatectomy in a Randomized Trial. PLoS One. 2015 Aug 28;10(8):e0135412. doi: 10.1371/journal.pone.0135412. eCollection 2015. PMID 26317357
- [Background] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097
- [Background] Barrio J, Errando CL, San Miguel G, Salas BI, Raga J, Carrion JL, Garcia-Ramon J, Gallego J. Effect of depth of neuromuscular blockade on the abdominal space during pneumoperitoneum establishment in laparoscopic surgery. J Clin Anesth. 2016 Nov;34:197-203. doi: 10.1016/j.jclinane.2016.04.017. Epub 2016 May 11. PMID 27687373
- [Background] Torensma B, Martini CH, Boon M, Olofsen E, In 't Veld B, Liem RS, Knook MT, Swank DJ, Dahan A. Deep Neuromuscular Block Improves Surgical Conditions during Bariatric Surgery and Reduces Postoperative Pain: A Randomized Double Blind Controlled Trial. PLoS One. 2016 Dec 9;11(12):e0167907. doi: 10.1371/journal.pone.0167907. eCollection 2016. PMID 27936214

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT05689957/Prot_SAP_ICF_000.pdf